CLINICAL TRIAL: NCT03431077
Title: An Open-Label, Multi-Center Study of LJPC-501 in Pediatric Patients Who Remain Hypotensive Despite Receiving Fluid Therapy and Vasopressor Therapy
Brief Title: A Study of LJPC-501 in Pediatric Patients With Hypotension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LJ501-CRH02
Record Dates: First submitted 2018-01-18; First posted 2018-02-13 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Catecholamine-resistant Hypotension (CRH); Distributive Shock; High Output Shock; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Angiotensin II; Giapreza

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LJPC-501 (Experimental): Angiotensin II administered via continuous infusion (1.25 - 40 ng/kg/min) for 24 hours up to 168 hours.
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II is a peptide hormone naturally produced by the body that regulates blood pressure via vasoconstriction and sodium reabsorption. LJPC-501 (angiotensin II) is being developed for the treatment of hypotension in patients who do not respond to fluids and vasopressor therapy.
  Other Names: Giapreza

SUMMARY:
The objective of this study is to evaluate the effect of LJPC-501 infusion on mean arterial pressure (MAP) or reduction in sum norepinephrine (NE) equivalent dosing, at Hour 2 after the start of LJPC-501, in pediatric patients who remain hypotensive despite receiving fluid therapy and vasopressor therapy. In addition, this study will evaluate the safety and tolerability of LJPC-501 in pediatric patients, the change in MAP over 24 hours after the start of LJPC-501, the change in serum lactate concentrations, and the change in Pediatric Logistic Organ Dysfunction (PELOD) scores.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients 2-17 years of age.
2. Patients requiring a total sum NE equivalent dose of > 0.1 μg/kg/min for a minimum of 2 hours and a maximum of 48 hours prior to initiation of LJPC-501 dosing.
3. Patients must have clinical diagnosis of distributive shock in the opinion of the treating team and the Investigator.
4. Patients are required to have central venous access, which is expected to remain present for the duration of LJPC-501 treatment.
5. Patients are required to have an indwelling arterial line, which is expected to remain present for at least the first 24 hours of LJPC-501 treatment.
6. Patients must have received at least 40 mL/kg of crystalloid or colloid equivalent over the initial 24-hour resuscitation period, and are adequately volume resuscitated in the opinion of the Investigator.
7. Parent or legal guardian is willing and able to provide informed consent and assist the patient in complying with all protocol requirements.

Exclusion Criteria:

1. Patients who are < 2 years of age or ≥ 18 years of age.
2. Patients with a standing Do Not Resuscitate order.
3. Patients diagnosed with acute occlusive coronary syndrome requiring pending intervention.
4. Patients on veno-arterial (VA) extracorporeal membrane oxygenation (ECMO).
5. Patients who have been on veno-venous (VV) ECMO for less than 6 hours.
6. Patients with a clinical suspicion of cardiogenic shock.
7. Patients who have a history of asthma or are currently experiencing bronchospasm requiring the use of inhaled bronchodilators and who are not mechanically ventilated.
8. Patients with acute mesenteric ischemia or a history of mesenteric ischemia.
9. Patients with active bleeding AND an anticipated need of multiple transfusions (within 48 hours of Screening).
10. Patients with active bleeding AND hemoglobin < 7 g/dL or any other condition that would contraindicate serial blood sampling.
11. Patients with an absolute neutrophil count (ANC) of < 500 cells/mm3.
12. Patients requiring more than 5 mg/kg daily of hydrocortisone or equivalent glucocorticoid medication as a standing dose.
13. Patients with an expected lifespan of < 12 hours or withdrawal of life support within 24 hours of Screening.
14. Patients with a known allergy to mannitol.
15. Patients who are currently participating in another investigational clinical trial.
16. Patients of childbearing potential who are known to be pregnant at the time of Screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-02-11 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
Effect of LJPC-501 on mean arterial pressure (MAP) | 2 hours
  To evaluate the effect of LJPC-501 infusion on mean arterial pressure (MAP).
Effect of LJPC-501 on sum norepinephrine (NE) equivalent dose | 2 hours
  To evaluate the effect of LJPC-501 in the reduction of the sum norepinephrine (NE) equivalent dosing.

SECONDARY OUTCOMES:
Effect of LJPC-501 on the incidence of treatment-emergent adverse events | Day 7
Effect of LJPC-501 on mean arterial pressure (MAP) | 24 hours
  To evaluate the change in MAP over 24 hours after the start of LJPC-501.
Effect of LJPC-501 on serum lactate | 2 hours and 24 hours
  To evaluate the change in serum lactate concentrations.
Effect of LJPC-501 on Pediatric Logistic Organ Dysfunction (PELOD) | 24 hours
  To evaluate change in Pediatric Logistic Organ Dysfunction (PELOD) score from Screening to 24 hours. The PELOD score is the sum of 6 individual item scores that totals 0-71 points. A higher PELOD score represents a worse outcome.
Effect of LJPC-501 on clinical chemistry laboratory parameters | 24 hours
  Safety data for clinical chemistry parameters including ALT, AST, ALP, total bilirubin, direct bilirubin, creatinine, BUN, phosphorus, glucose, albumin, calcium, bicarbonate, chloride, sodium, potassium, magnesium, PT, PTT, and INR. In addition, serum pregnancy test will be assessed at screening to confirm eligibility.
Effect of LJPC-501 on hematology laboratory parameters | 24 hours
  Safety data for laboratory hematology parameters including hemoglobin, hematocrit, platelets, and WBC.
Effect of LJPC-501 on blood pressure | Day 7
  Change in blood pressure (mmHg).
Effect of LJPC-501 on heart rate | Day 7
  Change in heart rate (bpm).
Effect of LJPC-501 on body temperature | Hour 24
  Change in body temperature (Celsius).
Effect of LJPC-501 on general health | Day 7
  Change in physical examination (by body system).
Effect of LJPC-501 on electrical activity of the heart | Hour 24
  Change in the electrical activity of the heart over a period of time using electrodes placed on the skin and recorded by electrocardiogram (ECG).
Effect of LJPC-501 on urine output | Day 7
  Change in urine output (ml).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigational Site, Charlotte, North Carolina
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, San Antonio, Texas